CLINICAL TRIAL: NCT06550869
Title: Application of Anterior Quadratus Lumborum Block at the Lateral Supra-arcuate Ligament Under Laparoscopic Direct Vision in Laparoscopic Renal Surgery：A Randomized, Controlled Trial
Brief Title: Application of Anterior Quadratus Lumborum Block at the Lateral Supra-arcuate Ligament Under Laparoscopic Direct Vision in Laparoscopic Renal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-0806
Record Dates: First submitted 2024-08-07; First posted 2024-08-13 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain; Analgesia; Quadratus Lumborum Block; Laparoscopic Renal Surgery
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLB-LSAL (Experimental): The patient received Anterior Quadratus Lumborum Block at the lateral supra-arcuate ligament under laparoscopic direct vision.
  Interventions: Procedure: Anterior Quadratus Lumborum Block at the lateral supra-arcuate ligament under laparoscopic direct vision
- LA (Active Comparator): The patient received local infiltration anesthesia.
  Interventions: Procedure: Local infiltration anesthesia

INTERVENTIONS:
Procedure: Anterior Quadratus Lumborum Block at the lateral supra-arcuate ligament under laparoscopic direct vision — The urologists find the inner arcuate ligament. The scalp needle is inserted from the midpoint of the lower edge of the inner or outer arcuate ligament towards the head to the dorsal side of the diaphragm. After withdrawing without blood, air, or cerebrospinal fluid, 2 ml of normal saline is first administered to observe the fluid spreading towards the head Then, 20 ml of 0.375% ropivacaine hydrochloride injection is administered.
  Arms: QLB-LSAL
Procedure: Local infiltration anesthesia — The urologists give local infiltration anesthesia with 20 ml of 0.375% ropivacaine hydrochloride injection.
  Arms: LA

SUMMARY:
Evaluation of the effectiveness of Anterior Quadratus Lumborum Block at the lateral supra-arcuate ligament under laparoscopic direct vision compared to local infiltration anesthesia for postoperative analgesia after laparoscopic renal surgery in patients.A randomized controlled trial involving 66 patients undergoing laparoscopic renal surgery will assign them randomly to an experimental group or a control group.The patients in experimental group will receive Anterior Quadratus Lumborum Block at the lateral supra-arcuate ligament under laparoscopic direct vision.The patients in control group will receive local infiltration anesthesia.The primary outcome measure is the cumulative consumption of intravenous morphine equivalents at postoperative 24 hours.The secondary outcomes include the cumulative consumption of intravenous morphine equivalents at postoperative 2, 4, 6, 12 and 48 hours, Numeric Rating Scale(NRS) score at rest and during activity (coughing) at postoperative 2, 6, 24 and 48 hours, Global Comfort Questionnaire(GCQ) Comfort Status Scale Score, Quality of Recovery-15(QoR-15) Postoperative Recovery Scale Score, time of the first press on the Patient-Controlled Analgesia pump, nausea, vomiting, skin itching, drowsiness, or other adverse reactions, regional anesthesia-related complications such as local anesthetic toxicity and length of postoperative hospital stay after surgery.

DETAILED DESCRIPTION:
The patients were 1:1 randomly assigned into groups by a clinical researcher not involved in the clinical procedures or data collection. The random numbers were generated by R studio 4.1.0 (R studio, Boston, MA, USA) software in a 1:1 ratio, with a block size of 8 for each group. The generated random numbers were sealed in opaque envelopes with sequential numbers. On the day of surgery, the envelope was opened by the protocol executor according to the recruitment order before the induction of general anesthesia.Data collection is in the charge of special personnel, and Case Report Form shall be filled in timely after data collection. At the same time, the electronic database was edited by Excel, and the electronic database was entered timely after filling in the paper Case Report form.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 80 years old;
* American Society of Anesthesiologists (ASA) physical status classification: I to III;
* Undergoing laparoscopic nephrectomy or partial nephrectomy (including robotic-assisted laparoscopic nephrectomy and partial nephrectomy).

Exclusion Criteria:

* Recent use of anticoagulant medications or abnormal coagulation function;
* Local infection at the puncture site or the presence of tumors, severe deformities, or systemic infection;
* Severe renal failure (serum creatinine > 442 μmol/L or requiring renal replacement therapy) or liver dysfunction (Child-Pugh Class C);
* Known allergy to local anesthetics or a family history of local anesthetic allergy;
* Preoperative cognitive impairment or inability to assess pain;
* Alcoholism, drug abuse, chronic opioid dependence, or the use of analgesics or psychotropic medications for more than 3 months;
* History of central and/or peripheral nervous system disorders or myasthenia gravis;
* Planned admission to the ICU;
* Surgical cancellation or patient refusal, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
intravenous morphine equivalents | Postoperative 24 hours
  The cumulative consumption of intravenous morphine equivalents

SECONDARY OUTCOMES:
intravenous morphine equivalents | Postoperative 2, 4, 6, 12 and 48 hours
  The cumulative consumption of intravenous morphine equivalents
Numeric Rating Scale | postoperative 2, 6, 24 and 48 hours
  Numeric Rating Scale（NRS） score at rest and during activity (coughing),the pain score is from 0-10,0 is no pain,10 is the most.
Global Comfort Questionnaire | Preoperative and postoperative 24 hours
  Global Comfort Questionnaire（GCQ） Kolcaba Scale Score,it includes 28 questions,1 is not agree with,4 is very agree with,the total score is 114.
Quality of Recovery-15 | Postoperative 24 hours
  Quality of Recovery-15（QoR-15） Postoperative Recovery Scale Score,it includes 15 questions,0 is the worst,10 is the best,total score is 150.
Time of the first press on Patient-Controlled Analgesia | Postoperative 48 hours
  Time of the first press on the Patient-Controlled Intravenous Analgesia pump
adverse reactions | Postoperative 72 hours
  Nausea, vomiting, skin itching, drowsiness, and other adverse reactions
Regional anesthesia-related complications | Postoperative 72 hours
  Regional anesthesia-related complications such as local anesthetic toxicity
Length of hospital stay | Postoperative 10 days
  Length of postoperative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Lina Yu, doctor, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Second affiliated Hospital School of Medicine,Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No